CLINICAL TRIAL: NCT06527222
Title: Ranolazine in ALS: Safety, and Effect on Cramps, Function and Quality of Life.
Brief Title: A Study of Ranolazine in ALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swathy Chandrashekhar, MBBS (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor-Investigator, Swathy Chandrashekhar, MBBS, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-43175
Record Dates: First submitted 2024-04-25; First posted 2024-07-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Motor Neuron Disease; Lou Gehrig's Disease; Placebo-Controlled
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ranolazine low dose (Experimental): Participants receive Ranolazine 500mg orally twice daily for 24 weeks.
  Interventions: Drug: Ranolazine
- Ranolazine high dose (Experimental): Participants receive Ranolazine 1000mg orally twice daily for 24 weeks.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Participants receive Ranolazine placebo orally twice daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — 500mg twice daily
  Other Names: Ranexa
  Arms: Ranolazine low dose
Drug: Ranolazine — 1000 mg twice daily
  Other Names: Ranexa
  Arms: Ranolazine high dose
Drug: Placebo — Ranolazine placebo twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, effect on cramps, function and quality of life of ranolazine versus placebo for the treatment of ALS.

DETAILED DESCRIPTION:
A prospective, multi center, double-blind, placebo-controlled, parallel group study of 2 doses of ranolazine (500 mg and 1000 mg twice daily) compared to placebo in patients with ALS.

Approximately 72 adults with ALS will be enrolled into the study in the United States at approximately 7 ALS treatment sites.

Participants will take oral ranolazine or placebo twice daily, attend a minimum of 5 onsite research visits, and 4 remote research visits.

The study is estimated to last 28 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with clinically definite, possible, probably, or lab-supported probable ALS per revised El Escorial criteria
* Breathing assessment called forced vital capacity (FVC) greater than or equal to 50%.
* Able to swallow pills at the start of the study and expected to for the length of the study.
* If on ALS modifying medications must be on a stable dose at least 30 days.
* Experiencing 4 or more cramps per week during a 2-week screening period.

Exclusion Criteria:

* Disease duration < 5 years
* Tracheostomy invasive ventilation, or noninvasive ventilation of more than 12 hours/day
* Pregnant or lactating, adults unable to consent, and prisoners
* Taking ranolazine or investigational drug or has received an investigational drug within 30 days (or 5 half-lives for drugs, whichever is longer) prior to screening
* Medically uncontrolled comorbidities (heart, liver, kidney disease)
* Baseline QTc interval prolongation >450 ms for men/ >470 ms for women, history of long QT syndrome, or medications which prolong the QT interval
* Participation in an experimental drug trial less than 30 days before screening
* Patients have to be on a stable dosage of any medications used to treat muscle cramps for ≥30 days or have been off these medications ≥30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Treatment-Emergent Adverse Events | Up to 28 weeks
  Patient report and medical records will be used to document adverse events and severe adverse events. Adverse events and severe adverse events will be assessed by the investigator and reported as needed for safety.
Tolerability of treatment assignment | Up to 28 weeks
  Tolerability will be measured by percentage of patients who complete the treatment assignment. Dose limiting toxicities will be determined by individual with an adverse event necessitating stopping.
Muscle cramp frequency | Up to 28 weeks
  Muscle cramp frequency will be measured numerically with a reporting period of 7 days.
  Changes will be compared from baseline to week 28 utilizing a modified Qualitative, Patient-Centered Assessment of Muscle Cramp Impact and Severity questionnaire.
Muscle cramp severity | Up to 28 weeks
  Muscle cramp severity will be measured by a score of 1-10 (1 being a very mild muscle cramp and 10 being the most severe cramp you ever experienced). Changes will be compared from baseline to week 28 utilizing a modified Qualitative, Patient-Centered Assessment of Muscle Cramp Impact and Severity questionnaire.
Muscle cramps impact on quality of life | Up to 28 weeks
  Effect of muscle cramps on quality of life will be measured with three patient reported yes or no questions (Yes indicating an impact on quality of life or no indicating no impact on quality of life). Changes will be compared from baseline to week 28 utilizing a modified Qualitative, Patient-Centered Assessment of Muscle Cramp Impact and Severity questionnaire
Safety Lab Cystatin C | Up to 28 weeks
  Patient safety measured with lab value Cystatin C in mg/L.
Safety Lab Estimated Glomerular Filtration Rate (eGFR) | Up to 28 weeks
  Patient safety measured with lab value eGFR in mL/min/1.73.
Safety Lab Alanine Transaminase (ALT) | Up to 28 weeks
  Patient safety measured with lab value ALT in IU/L.
Safety Lab Aspartate Transferase (AST) | Up to 28 weeks
  Patient safety measured with lab value AST in IU/L.
Safety Lab Alkaline Phosphatase (ALP) | Up to 28 weeks
  Patient safety measured with lab value ALP in IU/L.
Safety Lab Total Bilirubin | Up to 28 weeks
  Patient safety measured with lab value total bilirubin in mg/dL.

SECONDARY OUTCOMES:
Muscle strength | Up to 28 weeks
  Change in muscle strength over time as measured by hand grip and hand-held dynamometry (HHD) in pounds.
ALS Functional Rating Scale-Revised (ALSFRS-R) | Up to 28 weeks
  Change in disease severity over time as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R). Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Forced Vital Capacity (FVC) | Up to 28 weeks
  Change in respiratory function as measured by Forced Vital Capacity (FVC) in liters.
Serum neurofilament light | Up to 28 weeks
  Changes in serum neurofilament light measured from baseline to end of treatment assignment. Data will be collected to determine differences between placebo and Ranolazine treatment groups at completion of the study.
Lymphocyte Mitochondrial Function | Up to 28 weeks
  Change in mitochondrial function in lymphocytes measured from baseline to the end of treatment assignment. Data will be collected to determine differences between placebo and Ranolazine treatment groups at completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Statland, MD, Principal Investigator — University of Kansas Medical Center
Locations (7):
- United States (7):
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Kansas Medical Center: Wichita, Wichita, Kansas
  - University of Missouri Health Care, Columbia, Missouri
  - The Ohio State University, Columbus, Ohio
  - National Neuromuscular Research Institute, PLLC., Austin, Texas

IPD SHARING:
Plan to Share IPD: No